CLINICAL TRIAL: NCT06573762
Title: Remote Monitoring Using Commercially Available Activity Trackers and Computer Vision Provides a Holistic, Low-cost Assessment of Parkinson's Disease Symptoms
Brief Title: Home-Based Monitoring in Parkinson's Disease
Status: Recruiting | Type: Observational
Sponsor: Jacob E. Simmering (Other)
Responsible Party: Sponsor-Investigator, Jacob E. Simmering, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 202308199
Record Dates: First submitted 2024-08-21; First posted 2024-08-27 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Recently Referred for Possible Parkinson's Disease: Patients referred to the University of Iowa Hospitals and Clinics (UIHC) Movement Disorders Clinic for possible Parkinson's disease.
- Recently Diagnosed with Parkinson's Disease: Patients of the UIHC Movement Disorders Clinic with a recent (less than 6 months) diagnosis of Parkinson's disease.

SUMMARY:
The goal of this observational study is to learn about the usefulness of automated analysis of speech, physical activity measures tracked using wearable devices at home, and tremor detection measured using computer-vision analysis of smartphone video to detect impairments related to Parkinson's disease and improve prediction of one-year progression.

Participants will attend a short research visit at the University of Iowa. During this visit, they will make a video recording using a smartphone of them performing a fine motor task and audio recordings of pre-written text. They will be provided with an activity tracker and asked to wear it at home for four weeks. After four weeks, a video visit will be conducted and the speech and video tasks will be repeated.

DETAILED DESCRIPTION:
Two groups of participants will be recruited. Group 1 will be patients newly referred to the Movement Disorders clinic for evaluation of possible Parkinson's disease. Group 2 will be patients with a recent (within 6 months) diagnosis of Parkinson's disease.

Group 1 (Newly Referred) will attend a baseline visit where the following data will be collected:

* Unified Parkinson's Disease Rating Scale (UPDRS). The motor assessment tasks will be recorded using an iPad.
* Montreal Cognitive Assessment (MoCA).
* Cognitive function assessment using NIH Toolbox.
* Diagnosis made at the Movement Disorders Clinic (PD or not PD).
* SF-20 quality of life assessment. (Short Form 20)
* PDQ-39 quality-of-life assessment. (Parkinson's Disease Questionnaire 39)
* Tongue and lip strength using the Iowa Oral Pressure Instrument.
* Cognitive function assessment using NIH Toolbox.
* Audio recordings of:

  * Diadochokinesis (DDK) assessment.
  * Vowel prolongation assessment.
  * Sentence Intelligibility Test.
  * Reading the Grandfather, Bamboo, and Rainbow passages.
  * Recording of conversational speech.

Participants will be provided with an activity tracker and a research team member will help install any required apps on the participant's phone, configure and connect the activity tracker, provide a basic overview of how the app and tracker work, and answer any additional questions the participant may have.

The participant will then wear the activity tracker at home for 4 weeks. Text messages reminders will be sent following days with non-wear (no recorded heart rate or steps for multiple hours throughout the day) as a reminder to increase wear time.

At 4 weeks, the participant will complete a video visit using Microsoft Teams/Zoom with a study team member and the study participant. During the video visit, a recording of three different fine-motor skill tasks used in the UPDRS will be made. During the call, the study team member will provide coaching and direct the participant to repeat the audio and UPDRS fine motor task assessment at home while recording the video visit. At the end of the video visit, research team member will also collect questions about the ease and willingness to use the activity tracker and video call for disease monitoring and any open-ended comments the participant wishes to provide. This concludes the participants involvement in the study.

Group 2 (Recently Diagnosed) will attend a baseline visit where the following data will be collected:

* Unified Parkinson's Disease Rating Scale (UPDRS). The motor assessment tasks will be recorded using an iPad.
* Montreal Cognitive Assessment (MoCA).
* Cognitive function assessment using NIH Toolbox.
* Diagnosis made at the Movement Disorders Clinic (PD or not PD).
* SF-20 quality of life assessment.
* PDQ-39 quality-of-life assessment.
* Tongue and lip strength using the Iowa Oral Pressure Instrument.
* Cognitive function assessment using NIH Toolbox.
* Audio recordings of:

  * Diadochokinesis (DDK) assessment.
  * Vowel prolongation assessment.
  * Sentence Intelligibility Test.
  * Reading the Grandfather, Bamboo, and Rainbow passages.
  * Recording of conversational speech.

Participants will be provided with an activity tracker and a research team member will help install any required apps on the participant's phone, configure and connect the activity tracker, provide a basic overview of how the app and tracker work, and answer any additional questions the participant may have.

The participant will then wear the activity tracker at home for 4 weeks. Text messages reminders will be sent following days with non-wear (no recorded heart rate or steps for multiple hours throughout the day) as a reminder to increase wear time.

At 4 weeks, the participant will complete a video visit using Microsoft Teams/Zoom with a study team member and the study participant. During the video visit, a recording of three different fine-motor skill tasks used in the UPDRS will be made. During the call, the study team member will provide coaching and direct the participant to repeat the audio and UPDRS fine motor task assessment at home while recording the video visit. At the end of the video visit, research team member will also collect questions about the ease and willingness to use the activity tracker and video call for disease monitoring and any open-ended comments the participant wishes to provide.

At 11 months, the participant will be contacted to schedule a one-year research visit. Many patients return on 3-6 month intervals to the UIHC Movement Disorders Clinic and the research visit will ideally coordinate the participants routine visit for care.

At the one-year encounter, which will be an in-person research visit, the following data elements will be collected:

* Unified Parkinson's Disease Rating Scale (UPDRS).
* Montreal Cognitive Assessment (MoCA).
* Cognitive function assessment using NIH Toolbox.
* SF-20.
* PDQ-39 quality-of-life assessment.

Additionally, the research team will solicit any open-ended feedback the participant wants to share with the study team about their experience being in the study.

ELIGIBILITY:
Group 1: People newly referred with possible Parkinson's disease

Inclusion Criteria

1. Newly referred to UIHC Movement Disorders Clinic

Exclusion Criteria

1. Prior diagnosis of Parkinson's disease
2. Confined to wheelchair or bed
3. Non-English speaking
4. Prisoner status
5. Inability to provide own informed consent
6. Phone unable to support the Fitbit app

Group 2: People with a recent diagnosis of Parkinson's disease

Inclusion Criteria

1. Patient of UIHC Movement Disorders Clinic
2. Diagnosed with Parkinson's disease

Exclusion Criteria

1. First diagnosed > 6 months ago
2. Confined to wheelchair or bed
3. Non-English speaking
4. Prisoner status
5. Inability to provide own informed consent
6. Phone unable to support the Fitbit app

Ages: 50 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be drawn from the patients seen at the UIHC Movement Disorders Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with a Diagnosis of Parkinson's Disease | Baseline
  Among Group 1 (those newly referred to the clinic for possible Parkinson's disease), a primary outcome will be whether the diagnosis made by the provider in the clinic was Parkinson's disease versus any other diagnosis.
  This is not an outcome for Group 2 (those with a recent diagnosis of Parkinson's disease) as everyone in that group will have that diagnosis.
Change in Fine Motor Function | Baseline, One Year
  Motor function will be evaluated using the UPDRS rating system.
Change in Total Cognition Composite Function | Baseline, One Year
  Total Cognition Composite will be calculated using the NIH Toolbox Cognition Battery. This score has a range from 0 to 200 with healthy adults having a mean score of 100 with a standard deviation of 15. Higher scores are associated with better cognitive performance.
Change in Total Crystallized Cognition Function | Baseline, One Year
  Crystallized Cognition Composite will be calculated using the NIH Toolbox Cognition Battery. This score has a range from 0 to 200 with healthy adults having a mean score of 100 with a standard deviation of 15. Higher scores are associated with better cognitive performance.
Change in Total Fluid Cognition Function | Baseline, One Year
  Fluid Cognition Composite will be calculated using the NIH Toolbox Cognition Battery. This score has a range from 0 to 200 with healthy adults having a mean score of 100 with a standard deviation of 15. Higher scores are associated with better cognitive performance.
Change in Montreal Cognitive Assessment Scores | Baseline, One Year
  The Montreal Cognitive Assessment (MoCA) has a range of 0-30. Higher scores are associated with better cognitive function. Scores of 26 or higher are considered cognitively normal. Scores less than 26 are suggestive of cognitive impairment, with dementia scores being below 20 but without a universally-accepted cutoff.

SECONDARY OUTCOMES:
Change in Short Form Survey 20 (SF-20) Health Quality of Life | Baseline, One Year
  Health related quality of life will me measured using the Short Form Survey 20 (SF-20). SF-20 scores range from 0 to 100 with higher scores having greater quality-of-life.
Change in Parkinson's Disease Questionnaire 39 (PDQ-39) Quality of Life | Baseline, One Year
  Health related quality of life will me measured using the Parkinson's Disease Questionnaire 39 (PDQ-39). PDQ-39 scores range from 0 to 156 with lower scores reflecting less Parkinson's disease burden and higher scores associated with greater disease burden.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Simmering, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be deposited in the National Archive of Computerized Data on Aging (NACDA). Analytical code and documentation of study procedures will be shared both via the NACDA record and via GitHub repositories.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will be released to the broader research community when the paper dependent on those results is posted as a pre-print, published, or when the award period ends, whichever happens first.
Access Criteria: To access the data, researchers will use the standard processes at the NACDA to obtain access to the data. The data generated in this study will be suitable for public access as it will be deidentified. NACDA provides a brief data use agreement prohibiting redistribution, identifying participants, and requires citing the data resource. Access is granted through an NACDA account, which may be created through a Google, OrcID, or Facebook account.